CLINICAL TRIAL: NCT03198754
Title: Programmed Environmental Illumination (PEI) of Hospital Rooms to Prevent/Reduce Cancer-Related Fatigue During Hematopoetic Stem Cell Transplantation for Multiple Myeloma
Brief Title: Programmed Environmental Illumination (PEI) of Hospital Rooms to Prevent/Reduce Cancer-Related Fatigue
Acronym: PEI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, William H. Redd, Associated Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GCO 15-2009
Record Dates: First submitted 2017-06-21; First posted 2017-06-26 (Actual); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Cancer-related Problem/Condition; Depression; Circadian Rhythm Disorders
Keywords: Autologous Stem Cell Transplant; Multiple Myeloma; oncology; circadian rhythms; light therapy; Hematopoietic stem cell transplantation
MeSH Terms: conditions — Depression; Chronobiology Disorders; Multiple Myeloma; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Neither the study participant nor the research coordinator know that study condition of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PEI Experimental Light (Experimental): Ambient light fixture installed in the patient's hospital room
  Interventions: Device: PEI Experimental Light
- Comparison Light (Active Comparator): Ambient light fixture installed in the patient's hospital room
  Interventions: Device: Comparison Light

INTERVENTIONS:
Device: PEI Experimental Light — Ambient Light Fixture will turn on automatically and illuminate the hospital room from 7 to 10 AM each morning.
  Arms: PEI Experimental Light
Device: Comparison Light — Ambient Light Fixture will turn on automatically and illuminate the hospital room from 7 to 10 AM each morning.
  Arms: Comparison Light

SUMMARY:
A sample of 60 patients scheduled for HSCT in the treatment of MM will be recruited in the weeks to months prior to their hospitalization. Light therapy incorporating ambient Programmed Environmental Illumination (PEI) will be used in patient hospital rooms (during scheduled transplant) to control cancer-related fatigue (CRF). The FDA has certified that light therapy, like that used in this study, is a low-risk intervention. When admitted to the hospital for a stem cell transplant, there will be a light fixture in the hospital room which the researchers will be testing to see how it may affect cancer related fatigue, sleep quality, and other negative side effects often seen with the transplant and subsequent treatment. The light fixture will turn on and off by itself in the morning. There are two treatment arms used in the study, each of the arms uses different light intensities. The study treatment received, i.e. which of the two lights, will be chosen by chance, like flipping a coin. There is an equal chance of being given each study treatment. Participants will not be told which study treatment they are getting until after the study is completed. Each light will be turned on from 7 AM to 10AM every day during transplantation. While in the hospital, assessment of fatigue, sleep activity, depression, circadian rhythms, and quality of life will continue through the course of hospitalization (14-21 days of treatment, to determine immediate impact of sPI), then repeat at one month and three months post-discharge follow-ups (to determine lasting effects). Outcomes will be assessed through standardized scales (e.g., FACIT-Fatigue Scale) and objective measures (e.g., actigraphy, daysimeter for light monitoring, melatonin from urine collection, blood inflammatory markers, all explained below). This trial will: 1) be the first randomized clinical trial (RCT) to investigate the effects of sPI to prevent CRF and other biopsychosocial side effects of transplant; 2) focus on a distinct, relatively homogenous patient population (MM-HSCT patients) with high prevalence of CRF; and 3) explore possible circadian rhythm mediation via melatonin analysis and blood analysis. This investigation will have major public health relevance as it will determine if an inexpensive and low patient burden intervention (sPI) is able to control fatigue associated with medical illnesses and related problems.

ELIGIBILITY:
Inclusion Criteria:

* Who will undergo their first autologous HSCT procedure as treatment for multiple myeloma

AND:

* Who are currently 21 years of age or older
* English language proficient
* Able to provide informed consent

Exclusion Criteria:

* Under age 21
* Previous HSCT procedure (autologous or allogeneic)Pregnancy
* Eye Diseases which limit the ability of light to be processed (e.g., untreated cataracts, severe glaucoma, macular degeneration, blindness, pupil dilation problems or retina damage)
* Secondary cancer diagnosis within the last 5 years
* Severe sleep disorders (e.g., Narcolepsy)
* History of bipolar disorder or manic episodes (which is a contra-indication for light treatment)
* Severe psychological impairment (e.g., hospitalization for depressive episode in the past 12 months)
* Previous use of light therapy to alleviate fatigue or depressive symptoms

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William H. Redd, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Multiple Myeloma — https://ghr.nlm.nih.gov/condition/multiple-myeloma
- See also: Fatigue — https://medlineplus.gov/fatigue.html
- See also: Genetic and Rare Diseases Information Center — https://rarediseases.info.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 89 consented, but 16 not enrolled
Groups:
- Circadian Active Bright White Light (BWL): PEI Experimental Light: Ambient Light Fixture delivery of circadian active bright white light (BWL) installed in the patient's hospital room will turn on automatically and illuminate the hospital room from 7 to 10 AM each morning.
- Circadian Inactive Dim White Light (DWL): Comparison Light: Ambient Light Fixture delivery of circadian inactive dim white light (DWL) installed in the patient's hospital room will turn on automatically and illuminate the hospital room from 7 to 10 AM each morning.
Period: Overall Study
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Started | 38 | 35
Completed | 27 | 27
Not Completed | 11 | 8
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Lost to Follow-up | 4 | 3
Not completed — Ineligible | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL) | Total
Number analyzed (Participants) | 38 | 35 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.18 (8.507) | 58.58 (7.521) | 60.04 (8.083)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 24 | 22 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 8 | 22
  White | 24 | 21 | 45
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: FACIT-Fatigue Scale
Description: The FACIT-Fatigue scale is a13 item scale, full scale 0-52, with higher score indicating better functioning or less fatigue.
Time Frame: Baseline, Day 2, 7, 14, 28 and 90
Population: Data available only for participants who completed instrument for respective study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 38 | 35
score on a scale
  Baseline: number analyzed (Participants) | 38 | 33
  Baseline | 37.00 (9.80) | 35.06 (10.51)
  Day 2: number analyzed (Participants) | 31 | 29
  Day 2 | 38.71 (7.62) | 35.00 (11.32)
  Day 7: number analyzed (Participants) | 31 | 30
  Day 7 | 29.16 (11.32) | 26.37 (13.49)
  Day 14: number analyzed (Participants) | 30 | 31
  Day 14 | 35.97 (8.41) | 29.94 (13.59)
  Day 28: number analyzed (Participants) | 29 | 26
  Day 28 | 38.17 (11.26) | 35.46 (10.07)
  Day 90: number analyzed (Participants) | 23 | 22
  Day 90 | 42.30 (8.24) | 38.86 (9.49)

2. Secondary Outcome: Multidimensional Fatigue
Description: The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. Tested for its psychometric properties in cancer patients receiving radiotherapy, patients with the chronic fatigue syndrome, psychology students, medical students, army recruits and junior physicians, it was found to have good Test-retest Reliability (r=0.80) and great Internal Consistency (Cronbach's alpha = 0.92).
Time Frame: up to 3 months
Population: Instrument not used and data not collected.
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: The Pittsburgh Sleep Quality Index
Description: The Pittsburgh Sleep Quality Index consists of 19 self-rated instrument full scale from 0-21, with higher score indicating poorer sleep quality.
Time Frame: Baseline, Day 30 and Day 90
Population: Data available only for participants who completed instrument for respective study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 38 | 35
score on a scale
  Baseline: number analyzed (Participants) | 31 | 27
  Baseline | 6.03 (3.11) | 7.59 (4.58)
  Day 30 after discharge: number analyzed (Participants) | 24 | 24
  Day 30 after discharge | 5.79 (3.60) | 6.13 (2.82)
  Day 90 after discharge: number analyzed (Participants) | 20 | 20
  Day 90 after discharge | 4.80 (3.41) | 6.30 (3.74)

4. Secondary Outcome: SF-36 Scale
Description: Quality of life assessed using the SF-36 scale. The SF-36 is a multi-purpose, short form health survey consisting of 36 questions. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability
Time Frame: Baseline and 30 days post hospital discharge
Population: Data available only for participants who completed instrument for respective study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 15 | 13
score on a scale
  Emotional Well Being Scale Baseline | 76.000 (17.13393) | 75.3846 (19.83910)
  Emotional Well Being Scale Day 30 after discharge: number analyzed (Participants) | 6 | 5
  Emotional Well Being Scale Day 30 after discharge | 89.1667 (8.61201) | 76.0000 (16.35543)
  General Health Scale Baseline | 65.2778 (22.58508) | 52.8846 (17.95253)
  General Health Scale Day 30 after discharge: number analyzed (Participants) | 6 | 5
  General Health Scale Day 30 after discharge | 63.8889 (22.77100) | 58.3333 (27.63854)
  Physical Functioning Scale Baseline | 66.3333 (29.48769) | 64.4872 (30.49275)
  Physical Functioning Scale Day 30 after discharge: number analyzed (Participants) | 6 | 5
  Physical Functioning Scale Day 30 after discharge | 78.3333 (16.32993) | 75.0000 (23.97916)
  Limitations due to Physical Health Scale Baseline | 64.1667 (38.19787) | 55.6923 (30.74105)
  Physicial Limitations Scale Day30 after discharge: number analyzed (Participants) | 6 | 5
  Physicial Limitations Scale Day30 after discharge | 77.0833 (25.20747) | 77.5000 (25.61738)
  Energy Fatigue Scale Baseline | 63.3333 (11.77985) | 62.5000 (15.72882)
  Energy Fatigue Scale Day 30 after discharge: number analyzed (Participants) | 6 | 5
  Energy Fatigue Scale Day 30 after discharge | 69.7917 (15.52048) | 61.2500 (21.378)
  Pain Scale Baseline | 75.0000 (24.54951) | 59.6154 (29.82320)
  Pain Scale Day 30 after discharge: number analyzed (Participants) | 6 | 5
  Pain Scale Day 30 after discharge | 79.1667 (20.41241) | 72.5000 (28.50439)
  Limitations due to Emotional Problems Baseline | 86.1111 (29.49083) | 75.0000 (30.61862)
  Emotional Limitations Scale Day 30 after discharge: number analyzed (Participants) | 6 | 5
  Emotional Limitations Scale Day 30 after discharge | 83.3333 (30.27650) | 78.3333 (26.08746)
  Social Functioning Scale Baseline | 82.50000 (22.05917) | 75.9615 (19.40625)
  Social Functioning Scale Day 30 after discharge: number analyzed (Participants) | 6 | 5
  Social Functioning Scale Day 30 after discharge | 93.75000 (15.30931) | 85.0000 (16.29801)

5. Secondary Outcome: Number of Participants With Score 16 or Greater on CES-D (Center for Epidemiologic Studies Depression Scale)
Description: Number of participants with score 16 or greater on CES-D, 20 item questionnaire that reflects major dimensions of depression: depressed mood; feelings of guilt and worthlessness; feelings of helplessness and hopelessness; psychomotor retardation; loss of appetite; and sleep disturbance. Full score from 0- 20, with higher score indicating more symptomology.
Time Frame: Baseline, Day 2, Day 7, and Day 14 post transplant
Population: Data available only for participants who completed instrument for respective study visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 38 | 35
Participants
  baseline, prior to hospitalization: number analyzed (Participants) | 38 | 33
  baseline, prior to hospitalization | 10 | 11
  Day 2 post- transplant: number analyzed (Participants) | 31 | 29
  Day 2 post- transplant | 9 | 8
  Day 7, post-transplant: number analyzed (Participants) | 32 | 30
  Day 7, post-transplant | 13 | 15
  Day 14, post transplant: number analyzed (Participants) | 30 | 31
  Day 14, post transplant | 12 | 17

6. Secondary Outcome: CES-D (Center for Epidemiologic Studies Depression Scale)
Description: CES-D, 20 item questionnaire that reflects major dimensions of depression: depressed mood; feelings of guilt and worthlessness; feelings of helplessness and hopelessness; psychomotor retardation; loss of appetite; and sleep disturbance. Full score from 0- 20, with higher score indicating more symptomology.
Time Frame: Baseline, Day 2, 7, 14, 28, and 90
Population: Data available only for participants who completed instrument for respective study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 38 | 35
score on a scale
  baseline, prior to hospitalization: number analyzed (Participants) | 38 | 33
  baseline, prior to hospitalization | 11.00 (8.47) | 10.94 (8.12)
  Day 2: number analyzed (Participants) | 31 | 29
  Day 2 | 12.48 (9.64) | 12.48 (9.26)
  Day 7: number analyzed (Participants) | 32 | 30
  Day 7 | 15.13 (9.01) | 17.93 (11.16)
  Day 14: number analyzed (Participants) | 30 | 31
  Day 14 | 14.43 (8.78) | 18.58 (10.71)
  Day 28: number analyzed (Participants) | 28 | 26
  Day 28 | 9.75 (9.03) | 10.27 (7.94)
  Day 90: number analyzed (Participants) | 23 | 21
  Day 90 | 8.13 (7.41) | 6.95 (7.17)

7. Secondary Outcome: The Positive and Negative Affect Schedule (PANAS)
Description: PANAS is a 20-item self-report measure of positive and negative affect. Each item rated on a 5-point scale of 1 (not at all) to 5 (extremely), each subscale from 1-5, full score from 1-5, with higher score indicating more symptoms. Change in PANAS at Day 30 and Day 90 as compared to baseline.
Time Frame: Baseline, Day 30, Day 90
Population: Data available only for participants who completed instrument for respective study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 38 | 35
score on a scale
  PANAS Negative Baseline: number analyzed (Participants) | 22 | 19
  PANAS Negative Baseline | 1.6455 (.65154) | 1.9316 (.82060)
  PANAS Negative Day 30 after discharge: number analyzed (Participants) | 21 | 20
  PANAS Negative Day 30 after discharge | 1.6524 (.90312) | .93667 (1.5950)
  PANAS Negative Day 90 after discharge: number analyzed (Participants) | 21 | 24
  PANAS Negative Day 90 after discharge | 1.4333 (.70875) | 1.5417 (.90068)
  PANAS Positive Baseline: number analyzed (Participants) | 22 | 19
  PANAS Positive Baseline | 3.2475 (.98800) | 3.1351 (.92138)
  PANAS Positive Day 30 after discharge: number analyzed (Participants) | 21 | 20
  PANAS Positive Day 30 after discharge | 3.3238 (.99242) | 2.6850 (.96588)
  PANAS Positive Day 90 after discharge: number analyzed (Participants) | 21 | 24
  PANAS Positive Day 90 after discharge | 3.4778 (.94465) | 3.0208 (.89003)

8. Secondary Outcome: Change in Brief Symptoms Inventory-18 (BSI-18)
Description: Brief Symptom Inventory-18 (BSI-18) - self-report 18-item instrument. Raw scores on the BSI-18 are converted to t-scores based on gender-specific normative data from non-patient community dwelling U.S. adults. A T-score = 50 indicating average function compared to the reference population and a standard deviation of 10, with a higher score indicating more symptom.
Time Frame: Baseline and Day 90
Population: Thirty-eight participants were randomized to the bright white light condition (BWL) and 35 were randomized to the dim white light condition (DWL). Not all participants completed each measure at all time-points. For intent to treat analyses all participants need to be accounted for.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 38 | 35
T-score
  Baseline: number analyzed (Participants) | 16 | 17
  Baseline | .6560 (.49498) | .4714 (.61354)
  Day 90: number analyzed (Participants) | 21 | 22
  Day 90 | .3280 (.48206) | .3763 (.67975)

9. Secondary Outcome: Fatigue Line Scale
Description: Simple numeric graphic rating scale, marked on a line numbering 0-100, with higher score indicating more fatigue. Replaces the FACIT fatigue scale for daily fatigue assessment during inpatient procedures.
Time Frame: baseline, day 2, 7, and 14
Population: Data available only for participants who completed instrument for respective study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 38 | 35
score on a scale
  Baseline: number analyzed (Participants) | 34 | 28
  Baseline | 34.62 (26.41) | 33.04 (23.35)
  Day 2: number analyzed (Participants) | 33 | 28
  Day 2 | 40.21 (24.19) | 33.21 (21.14)
  Day 7: number analyzed (Participants) | 33 | 28
  Day 7 | 55.55 (28.45) | 52.86 (27.16)
  Day 14: number analyzed (Participants) | 17 | 13
  Day 14 | 47.65 (21.59) | 44.23 (33.22)

10. Secondary Outcome: Multidimensional Fatigue Symptom Inventory- Short Form (MFSI-SF)
Description: Multidimensional Fatigue Symptom Inventory- Short Form (MFSI-SF) is a 30-item short form of the MFSI that measures ﬁve dimensions: general, physical, emotional, mental fatigue, and vigor. Each item is rated on a ﬁve-point Likert scale from 0 (not at all) to 4 (extremely). The total MFSI-SF score ranges from 0-4, with a higher score indicating a higher fatigue level.
Time Frame: Baseline, Day 30 after Discharge, Day 90 after Discharge
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 38 | 35
score on a scale
  Baseline: number analyzed (Participants) | 22 | 19
  Baseline | 3.1689 (2.77373) | 3.0368 (2.18310)
  Day 30 after Discharge: number analyzed (Participants) | 21 | 19
  Day 30 after Discharge | 2.2365 (2.02204) | 2.8088 (2.30284)
  Day 90 after Discharge: number analyzed (Participants) | 21 | 22
  Day 90 after Discharge | 2.2093 (1.75925) | 2.2371 (2.65162)

11. Secondary Outcome: Sleep Latency
Description: Sleep latency measured by actigraph - Sleep latency is the average period of time between bed time and sleep start time
Time Frame: Baseline, Day 2, Day 7, 3rd day post Engraftment, Discharge
Population: Data available only for participants who completed instrument for respective study visits.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 27 | 27
minutes
  Baseline: number analyzed (Participants) | 23 | 27
  Baseline | 6.1739 (7.61370) | 12.1481 (23.62154)
  Day 2: number analyzed (Participants) | 20 | 26
  Day 2 | 4.3000 (8.90949) | 9.1538 (14.94173)
  Day 7: number analyzed (Participants) | 20 | 27
  Day 7 | 6.8500 (6.25153) | 4.7778 (6.81251)
  3rd day post Engraftment: number analyzed (Participants) | 16 | 22
  3rd day post Engraftment | 7.1875 (10.88252) | 4.0909 (4.92718)
  Discharge, average 14 days: number analyzed (Participants) | 16 | 19
  Discharge, average 14 days | 3.1250 (5.40216) | 6.1579 (7.55912)

12. Secondary Outcome: Sleep Efficiency
Description: Sleep efficiency measured by actigraph - Sleep efficiency is defined as the average percentage of time in bed actually spent sleeping
Time Frame: Baseline, Day 2, Day 7, 3rd day post Engraftment, Discharge
Population: Data available only for participants who completed instrument for respective study visits.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 27 | 27
percentage of time
  Baseline: number analyzed (Participants) | 23 | 27
  Baseline | 88.1517 (12.11416) | 89.3481 (6.34251)
  Day 2: number analyzed (Participants) | 20 | 26
  Day 2 | 87.3555 (8.01844) | 86.4504 (10.24487)
  Day 7: number analyzed (Participants) | 20 | 27
  Day 7 | 86.2340 (7.27702) | 86.3233 (9.42600)
  3rd day post Engraftment: number analyzed (Participants) | 16 | 22
  3rd day post Engraftment | 84.5994 (7.92472) | 83.0605 (13.49365)
  Discharge, average 14 days: number analyzed (Participants) | 16 | 19
  Discharge, average 14 days | 85.1650 (7.88246) | 84.5600 (12.06957)

13. Secondary Outcome: Wake Time
Description: Wake time measured by actigraph. Wake time is the average number of minutes the participant spent awake each night during the 5 day period. Baseline assessments were taken before transplant and day 2 is two days after transplant which is at least one week after the baseline.
Time Frame: Baseline, Day 2, Day 7, 3rd day post Engraftment, Discharge
Population: Data available only for participants who completed instrument for respective study visits.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 27 | 27
minutes
  Baseline: number analyzed (Participants) | 23 | 27
  Baseline | 41.7391 (50.64602) | 40.5556 (37.40561)
  Day 2: number analyzed (Participants) | 20 | 26
  Day 2 | 56.1000 (40.07743) | 57.2308 (44.75382)
  Day 7: number analyzed (Participants) | 20 | 27
  Day 7 | 57.6000 (42.40209) | 69.0370 (57.24675)
  3rd day post Engraftment: number analyzed (Participants) | 16 | 22
  3rd day post Engraftment | 68.1250 (35.86805) | 84.6364 (88.30981)
  Discharge, average 14 days: number analyzed (Participants) | 16 | 19
  Discharge, average 14 days | 62.6875 (33.40802) | 63.3158 (57.05363)

14. Secondary Outcome: Wake Percent
Description: Wake percent measured by actigraph - Wake percent is the average percent of each night spent awake
Time Frame: Baseline, Day 2, Day 7, 3rd day post Engraftment, Discharge
Population: Data available only for participants who completed instrument for respective study visits.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 27 | 27
percentage of time
  Baseline: number analyzed (Participants) | 23 | 27
  Baseline | 9.4665 (11.90539) | 7.9574 (6.25857)
  Day 2: number analyzed (Participants) | 20 | 26
  Day 2 | 11.5900 (7.51981) | 11.0746 (7.82651)
  Day 7: number analyzed (Participants) | 20 | 27
  Day 7 | 11.9765 (7.21864) | 12.3589 (9.11993)
  3rd day post Engraftment: number analyzed (Participants) | 16 | 22
  3rd day post Engraftment | 13.1819 (6.67063) | 15.7973 (13.55268)
  Discharge, average 14 days: number analyzed (Participants) | 16 | 19
  Discharge, average 14 days | 12.6494 (6.22923) | 13.0326 (9.44681)

15. Secondary Outcome: Sleep Time
Description: Sleep time measured by actigraph. Sleep time - average number of minutes the participant was asleep each night during the 5 day period. Baseline assessments were taken before transplant and day 2 is two days after transplant which is at least one week after the baseline.
Time Frame: Baseline, Day 2, Day 7, 3rd day post Engraftment, Discharge
Population: Data available only for participants who completed instrument for respective study visits.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 27 | 27
minutes
  Baseline: number analyzed (Participants) | 23 | 27
  Baseline | 396.0000 (106.94731) | 444.2407 (120.45869)
  Day 2: number analyzed (Participants) | 20 | 26
  Day 2 | 423.3500 (102.93753) | 458.3077 (122.00419)
  Day 7: number analyzed (Participants) | 20 | 27
  Day 7 | 422.9500 (124.38246) | 469.0370 (103.74839)
  3rd day post Engraftment: number analyzed (Participants) | 16 | 22
  3rd day post Engraftment | 445.0000 (114.98870) | 412.9545 (103.99472)
  Discharge, average 14 days: number analyzed (Participants) | 16 | 19
  Discharge, average 14 days | 442.7500 (139.03261) | 429.0526 (142.22223)

16. Secondary Outcome: Sleep Percent
Description: Sleep percent measured by actigraph. Sleep percent is the percent of time spent in bed that the participant is asleep.
Time Frame: Baseline, Day 2, Day 7, 3rd day post Engraftment, Discharge
Population: Data available only for participants who completed instrument for respective study visits.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 27 | 27
percentage of time
  Baseline: number analyzed (Participants) | 23 | 27
  Baseline | 90.5335 (11.90539) | 92.0426 (6.25857)
  Day 2: number analyzed (Participants) | 20 | 26
  Day 2 | 88.4100 (7.51981) | 88.9254 (7.82651)
  Day 7: number analyzed (Participants) | 20 | 22
  Day 7 | 88.0265 (7.21864) | 87.6411 (9.11993)
  3rd day post Engraftment: number analyzed (Participants) | 16 | 22
  3rd day post Engraftment | 86.8181 (6.67063) | 84.2027 (13.55268)
  Discharge, average 14 days: number analyzed (Participants) | 16 | 19
  Discharge, average 14 days | 87.3506 (6.22923) | 86.9674 (9.44681)

17. Secondary Outcome: Melatonin
Description: Melatonin level
Time Frame: Baseline and Discharge
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
Number analyzed (Participants) | 27 | 27
ng/ml
  Baseline | 21.5116 (20.83586) | 41.2025 (64.54599)
  Discharge, average 14 days | 31.6728 (45.04760) | 19.0317 (23.11714)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Circadian Active Bright White Light (BWL) | Circadian Inactive Dim White Light (DWL)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/35
Other Adverse Events (participants affected / at risk) | 0/38 | 0/35

LIMITATIONS AND CAVEATS:
Relatively small sample size and did not include post-hospitalization assessments of depressive symptoms. Third, the potential mechanisms underlying the effects of BWL on depressive symptoms were not examined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03198754/Prot_SAP_000.pdf